CLINICAL TRIAL: NCT03439410
Title: Development of a Mathematical Model of Clinical Complexity and of an Index for Its Practical Evaluation in Observational Prospective Longitudinal Studies. San MAtteo Complexity Study
Brief Title: Clinical Complexity in Internal Medicine Wards. San MAtteo Complexity Study
Acronym: SMAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Gino Roberto Corazza, Full Professor of Internal Medicine, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: SMAC Study
Record Dates: First submitted 2018-02-06; First posted 2018-02-20 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Multimorbidity; Health Knowledge, Attitudes, Practice
Keywords: Internal medicine; Chronic disease; Healthcare expenditure
MeSH Terms: conditions — Behavior; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Internal Medicine ward: The Clinical Complexity Index (CCI) will be administered to all patients admitted to the ward.
  Interventions: Other: Clinical Complexity Index
- Subacute ward: The Clinical Complexity Index (CCI) will be administered to all patients admitted to the ward.
  Interventions: Other: Clinical Complexity Index

INTERVENTIONS:
Other: Clinical Complexity Index — Clinical Complexity Index (CCI) will be administered at the time of admission to the ward.

SUMMARY:
The progressive rising of multimorbidity, which has been always considered the hallmark of clinical complexity (CC), has made management of the "complex" patient one of the most topical and challenging issues in medicine. However, patient-related factors (multimorbidity, age, frailty, disease severity) pertain only to the biological complexity, while CC is the result of the dynamic interaction between biological complexity and a number of other coexisting factors (socio-economic, cultural, behavioural, environmental). Starting from these premises, the investigators designed a five-year observational prospective longitudinal study that aims to validate and compare a CC score system on a large cohort of patients (n=1000) admitted in internal medicine wards. Clinicians, biostatisticians and epidemiologists will cooperate into the project. A questionnaire that encompasses the main biological and extra-biological factors was designed (Clinical Complexity Index, CCI) by a multiprofessional consensus. This questionnaire will be administered by the investigators to the patients and validated. Consecutive patients will be enrolled every other week for two years and followed-up for 5 years. The primary endpoint will be the validation of the CCI. Thereafter, the investigators will evaluate the correlation between the CCI and the length of stay of the index hospitalization, assuming that a higher CCI score is associated with longer length of stay. The secondary endpoints will be the demonstration of the association between higher CCI score and more health resources utilization (i.e., evaluating occurrence of hospital readmissions, number of accesses to the emergency room, visits at the outpatient clinic, different drugs prescribed and hospital reimbursement according to the local diagnosis-related group [DRG] system) along with worse prognosis (mortality at 1 and 5 years).

DETAILED DESCRIPTION:
The Clinical Complexity Index (CCI) that will be validated is made of 25 different variables, divided into 5 domains (biological, socioeconomic, behavioral, environmental, cultural). All variables were dichotomised and were coded -1 (absence of the variable) and +1 (presence of the variable). For each variable, the answer "yes" increases the degree of complexity. See Citations for further details.

Here is the CCI that will be used in the study:

BIOLOGICAL DOMAIN Age > 75 years yes☐ +1 no☐ -1 Intake ≥ 5 medications yes☐ +1 no☐ -1 Cumulative Illness Rating Scale (CIRS) > 3 and/or CIRS severity >3 yes☐ +1 no☐ -1 ↑ frailty (Edmonton Frail Scale > 5) yes☐ +1 no☐ -1

↓ mobilization (Barthel<60) yes☐ +1 no☐ -1

SOCIO-ECONOMIC DOMAIN Living alone yes☐ +1 no☐ -1 Income < 1000 €/month yes☐ +1 no☐ -1 Unemployment/precarious work yes☐ +1 no☐ -1 Dependent/disabled family member yes☐ +1 no☐ -1 Need for a caregiver yes☐ +1 no☐ -1

BEHAVIOURAL DOMAIN Inadequate adherence to medications yes☐ +1 no☐ -1 Active smoking of at least 4 cigarettes/day yes☐ +1 no☐ -1 Alcohol (>3 Alcohol Units/day) and/or drug abuse yes☐ +1 no☐ -1 Inappropriate diet yes☐ +1 no☐ -1 Cognitive impairment (Short Blessed Test > 9) yes☐ +1 no☐ -1

ENVIRONMENTAL DOMAIN Institutionalization yes☐ +1 no☐ -1 Difficult access to healthcare yes☐ +1 no☐ -1 Presence of home architectural barriers yes☐ +1 no☐ -1 Occupational exposure to toxins yes☐ +1 no☐ -1 Air pollution yes☐ +1 no☐ -1

CULTURAL DOMAIN Schooling < 8 years yes☐ +1 no☐ -1 Insufficient access to information yes☐ +1 no☐ -1 Lack of adherence to health screening programs yes☐ +1 no☐ -1 Language barriers yes☐ +1 no☐ -1 Perceived discrimination yes☐ +1 no☐ -1

The investigators will administer the CCI to all patients admitted to the wards (Internal Medicine and Subacute ward), according the study protocol. All the enrolled patients will be followed-up with a phone call after after discharge (at 4-8-12 months) for collecting the following data: occurrence of hospital readmission within 1 month after discharge; the number of readmissions; the number of accesses to the emergency room (ER); the number of visits at the outpatient clinic; the number of different drugs prescribed; mortality. Mortality will also be assessed once a year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Hospitalized in one of the participating Units (Internal Medicine wards or Subacute ward)

Exclusion Criteria:

* Already enrolled in the study during a previous hospitalization
* Denied informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the aforementioned wards will be enrolled in the study during the time of the study
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-11-06 (Estimated); Study Completion 2022-11-06 (Estimated)

PRIMARY OUTCOMES:
Validation of the Clinical Complexity Index (CCI) | 2 years
  Validation of the Clinical Complexity Index (CCI) proposed in the project (see first Citation and Study Description for further details). This index should measure patients' clinical complexity, including biological, socioeconomic, cultural, behavioral, and envirnomental domains. The total score range is -25 to +25 (-5 to +5 per each domain). The investigators expect that a higher value is associated with a worse outcome (higher clinical complexity).

SECONDARY OUTCOMES:
Length of stay | 2 years
  The investigators will measure the length of stay (unit of measurement: days) of each enrolled patient.
Healthcare expenditure and utilization | 1 year
  To demonstrate the association of the Clinical Complexity Index (CCI) with the use of health resources, including the occurrence of hospital readmission within 1 month; the number of readmissions during the first 12 months; the number of accesses to the emergency room (ER) during the first 12 months; the number of visits at the outpatient clinic during the first 12 months; the number of different drugs prescribed during the first 12 months; the hospital reimbursement according to the Regional DRG system for the index hospitalization. Each of these items will be separately analyzed.
Mortality | 5 years
  To evaluate the association between a higher Clinical Complexity Index (CCI) score and mortality at 1 and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Gino R Corazza, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD), anonymized and aggregated, that underlie results in a publication.
Supporting Information: SAP, CSR
Time Frame: Only on future articles that will be published.

REFERENCES:
- [Background] Palese A, Brusaferro S. A multidimensional vector model measuring clinical complexity may increase effectiveness in patient assessment. Intern Emerg Med. 2017 Dec;12(8):1287-1289. doi: 10.1007/s11739-017-1722-9. Epub 2017 Aug 4. No abstract available. PMID 28779449
- [Result] Corazza GR, Klersy C, Formagnana P, Lenti MV, Padula D; Consensus Panel. A consensus for the development of a vector model to assess clinical complexity. Intern Emerg Med. 2017 Dec;12(8):1313-1318. doi: 10.1007/s11739-017-1709-6. Epub 2017 Jul 14. PMID 28710713
- [Derived] Lenti MV, Brera AS, Ballesio A, Croce G, Padovini L, Bertolino G, Di Sabatino A, Klersy C, Corazza GR. Resilience is associated with frailty and older age in hospitalised patients. BMC Geriatr. 2022 Jul 10;22(1):569. doi: 10.1186/s12877-022-03251-9. PMID 35818046